CLINICAL TRIAL: NCT02513199
Title: Assessment of Response of Unresectable Hepatocellular Carcinoma to Combination Chemoembolization and Stereotactic Body Radiation Therapy
Brief Title: Combination Chemoembolization and Stereotactic Body Radiation Therapy in Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Michael Buckstein, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1671
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Trans-Arterial Chemoembolization; Stereotactic Body Radiation Therapy; HCC; TACE; SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with HCC (Experimental): Participants with HCC with a lesion greater than 3 cm treated with TACE/SBRT combination
  Interventions: Radiation: SBRT; Drug: TACE

INTERVENTIONS:
Radiation: SBRT — Radiation is to be delivered to 30-45 Gy in 5 fractions. 40 Gy in 5 fractions will be utilized, unless dose constraints preclude it. Treatment will optimally be delivered every other day with no more than 3 fractions per week. The ideal treatment team will be less than 15 total days.
  Other Names: Stereotactic Body Radiation Therapy
Drug: TACE — two sessions of standard TACE with ethiodol separated by a 4-week interval.
  Other Names: Trans-Arterial Chemoembolization

SUMMARY:
The purpose of this study is to develop better ways to treat liver cancer, known as hepatocellular carcinoma or HCC, while it is still in the liver. Many treatments exist to treat tumors in the liver when they are small but after they grow past a certain size, local therapies such as surgery, Trans-Arterial Chemo Embolization (TACE), or Radiofrequency Ablation (RFA) are not effective. The purpose of this study to test the combination of two known treatments - TACE and Stereotactic Body Radiation Therapy (SBRT) - to be used together to treat larger or difficult to access liver tumors. Each treatment has been shown to work well but has limitations. The study will combine the treatments in an organized sequence and monitor closely how effective this combination controls tumors.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third ranked cause of global cancer mortality. There is an increasing incidence of HCC in the United States over the last twenty years, largely due to the Hepatitis C epidemic but increasingly related as well to nonalcoholic fatty liver disease.

This is a non-randomized pilot study to assess the objective response rate and durability of response of combination Trans-Arterial Chemoembolization (TACE) with immediate stereotactic body radiation therapy (SBRT) in the treatment of unresectable hepatocellular carcinoma (HCC). Eligible patients will be selected based on having a lesion greater than 3 cm which would make them ineligible for other local therapies such as TACE and thermal ablation (TA). Eligible, consented, and registered patients will be treated with two sessions of standard TACE with ethiodol separated by a 4-week interval. After ensuring adequate return to baseline liver function, the patients will then be treated with SBRT to the targeted lesion to 30-45 Gy in 5 fractions. Tumor response will be assessed using mRECIST criteria as well diffusion weight imaging (DWI) via Magnetic Resonance Imaging (MRI) surveillance. In addition, tolerability and toxicity will be recorded via CTCAE v. 4.0. The essential hypothesis of this study is that combination TACE and SBRT for > 3 cm HCC will produce higher response rates and durable control compared to TACE alone.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with HCC either pathologically or by the American Association for the Study of Liver Diseases (AASLD) radiographic criteria (Bruix Hepatology 2011). The criteria specifies CT or MRI intense arterial uptake followed by "washout" of contrast in the venous-delayed phases. Any atypical lesions must be confirmed by biopsy.
* A single liver lesion with tumor size ≥ 3 cm as defined as maximal diameter in the axial dimension on MRI. Included in the measurement are both enhancing and non-enhancing components of the lesion.
* Maximum tumor size of 7 cm as defined as maximal diameter in the axial dimension on MRI.
* Age ≥ 18 years
* Child-Pugh class A or B7 without ascites
* ECOG score 0
* No prior treatment of current HCC. However, recurrent HCC after resection may be included.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnancy which will be assessed via pregnancy test prior to TACE and repeated prior to SBRT.
* Metastatic disease outside of the liver
* Vascular invasion as evidenced by vessel occlusion or radiographic evidence of tumor thrombus.
* Contraindications to MRI, including claustrophobia, metallic implants, and pacemakers
* Tumor for which adequate radiation dosage cannot be safely delivered (see dose constraints below)
* Prior therapeutic radiation therapy to the abdomen and/or lower thorax as defined as below the carina to the pelvic inlet.
* Inability to provide informed consent based on persistent lack of understanding, inability to find adequate translation, impaired mental status such as mental retardation, drug induced, or traumatic brain injury.
* Multiple liver tumors making the patient a BCLC Stage B
* Prior treatment, except for surgical resection, to the lesion being targeted in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Buckstein, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Buckstein M, Kim E, Ozbek U, Tabrizian P, Gunasekaran G, Facciuto M, Rosenzweig K, Llovet JM, Schwartz M. Combination Transarterial Chemoembolization and Stereotactic Body Radiation Therapy for Unresectable Single Large Hepatocellular Carcinoma: Results From a Prospective Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2022 Oct 1;114(2):221-230. doi: 10.1016/j.ijrobp.2022.05.021. Epub 2022 May 26. PMID 35643250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2014 and 2020, of 33 potential candidates screened at the Liver Cancer Program at Mount Sinai Hospital in New York, NY, 32 patients were finally enrolled in the study.
Groups:
- TACE/SBRT Combination: Participants with HCC with a lesion greater than 3 cm treated with TACE/SBRT combination.
  SBRT: Radiation is to be delivered to 30-45 Gy in 5 fractions. 40 Gy in 5 fractions will be utilized, unless dose constraints preclude it. Treatment will optimally be delivered every other day with no more than 3 fractions per week. The ideal treatment team will be less than 15 total days.
  TACE: two sessions of standard TACE with ethiodol separated by a 4-week interval.
Period: Treatment
Arm/Group | TACE/SBRT Combination
Started | 32
Completed | 30
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Period: Follow-Up
Arm/Group | TACE/SBRT Combination
Started | 30
Completed | 19
Not Completed | 11
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 67.5 [52 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of participants with HCV Etiology [Count of Participants; unit: Participants] — Number of participants with Hepatitis C Virus (HCV) Etiology
  Participants | 21
Number of Participants with HBV Etiology [Count of Participants; unit: Participants] — Number of Participants with Hepatitis B Virus (HBV) Etiology
  Participants | 3
Number of Participants with NASH Etiology [Count of Participants; unit: Participants] — Number of Participant with NASH - Nonalcoholic Steatohepatitis Etiology of HCC
  Participants | 3
Number of Participants with Alcohol Etiology for HCC [Count of Participants; unit: Participants] | 4
Child-Turcotte-Pugh (CTP) Score [Count of Participants; unit: Participants] — Class A - 5 to 6 points, least severe liver disease, one- to five-year survival rate: 95 percent
  Class B - 7 to 9 points, moderately severe liver disease, one- to five-year survival rate: 75 percent
  Class C - 10 to 15 points, most severe liver disease, one- to five-year survival rate: 50 percent
  Higher score indicates more severe
  Participants
    A5 | 18
    A6 | 10
    B7 or greater | 2
Albumin-Bilirubin (ALBI) Grade [Count of Participants; unit: Participants] — Grade 1 - ALBI ≤-2.60
  Grade 2 - ALBI >-2.60 to ≤-1.39
  Grade 3 - ALBI >-1.39
  Higher grade indicates poorer health outcomes
  Participants
    Grade 1 | 15
    Grade 2 | 16
    Grade 3 | 1
ALBI Score [Median (Full Range); unit: ALBI score] — ALBI score = (log10 bilirubin [µmol/L] × 0.66) + (albumin [g/L] × - 0.085)^9
  Higher score indicates poorer health.
  ALBI score | -2.45 [-3.47 to 1.03]
Platelet Count [Median (Inter-Quartile Range); unit: 10^3 cells/uL] | 150 [56 to 365]
Tumor Size [Median (Full Range); unit: cm] | 4.6 [4 to 6.9]
Number of Participants with Tumor Size ≥5 [Count of Participants; unit: Participants] | 12
Alpha-fetoprotein (AFP) [Median (Full Range); unit: ng/mL] | 7.9 [2 to 7141]
Number of Participants with AFP ≥400ng/mL [Count of Participants; unit: Participants] | 5
Tumor Dose [Median (Full Range); unit: Gy] | 45 [30 to 50]
Biologic Effective Dose [Median (Inter-Quartile Range); unit: Gy] | 86 [48 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Rate
Description: Tumor response will be assessed using mRECIST criteria as well diffusion weight imaging (DWI) via Magnetic Resonance Imaging (MRI) surveillance.
  * Complete response (CR): Disappearance of all target lesions
  * Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
  * Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: up to 72 months
Measure: Count of Participants; unit: Participants
Groups:
- TACE/SBRT Combination: SBRT: Radiation is to be delivered to 30-45 Gy in 5 fractions. 40 Gy in 5 fractions will be utilized, unless dose constraints preclude it. Treatment will optimally be delivered every other day with no more than 3 fractions per week. The ideal treatment team will be less than 15 total days.
  TACE: two sessions of standard TACE with ethiodol separated by a 4-week interval.
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 30
Participants
  Complete response (CR) | 20
  Partial response (PR) | 9
  Stable disease (SD) | 0
  Progressive disease (PD) | 1

2. Secondary Outcome: Time to CR
Description: Time to Complete Remission (CR)
Time Frame: up to 72 months
Measure: Median (Full Range); unit: months
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 30
months | 10.1 [1 to 72]

3. Secondary Outcome: Time to Progression (TTP)
Description: The time to progression of the treated lesion. Median TTP, as defined as progression events (not including death), was not reached because 50% of events were not achieved. Because a sufficient number of progression events did not happen at the time of study censure, a median could not be reported. Therefore, mean is reported which can be reported irrespective of events.
Time Frame: up to 80 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 30
months | 76.60 (23.40)

4. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: The overall survival as defined from completion of treatment until death
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 32
Participants | 20

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS), defined as time between enrollment and tumor progression assessed by mRECIST or death, local control (LC), and toxic effects. LC was defined as either absence of radiographic progression or a secondary intervention (ie, surgery or TACE) made to the index lesion due to a perceived incomplete treatment response.
Time Frame: up to 72 months
Population: under efficacy, median PFS 35 months. under conclusions, PFS median 2.9 years (34.8months) and later on says PFS was 13.9 months
Measure: Median (Full Range); unit: months
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 30
months | 35 [15 to 72]

6. Secondary Outcome: Change in Child-Turcotte-Pugh (CTP) Score
Description: Overall rate of toxic effects as measured by change in Child-Turcotte-Pugh (CTP) score at 3 months as compared to baseline.
  The Child-Turcotte-Pugh (CTP) is a scale that assesses a patients baseline liver function and can help predict morbidity and mortality based on that score.
  Class A - 5 to 6 points, least severe liver disease, one- to five-year survival rate: 95 percent
  Class B - 7 to 9 points, moderately severe liver disease, one- to five-year survival rate: 75 percent
  Class C - 10 to 15 points, most severe liver disease, one- to five-year survival rate: 50 percent
  Higher scores correlate with more general mortality.
Time Frame: 3 months
Population: one participant did not have pre and post-CTP scores.
Measure: Count of Participants; unit: Participants
Arm/Group | TACE/SBRT Combination
Number analyzed (Participants) | 29
Participants
  Increase | 3
  Decrease | 3
  No Change | 22
  Decompensated | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | TACE/SBRT Combination
All-Cause Mortality (participants affected / at risk) | 12/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT02513199/Prot_SAP_000.pdf